CLINICAL TRIAL: NCT00418431
Title: Intravitreal Bevacizumab for the Treatment of Central Serous Chorioretinopathy
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-0016
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

INTERVENTIONS:
Drug: Intravitreal injection of Bevacizumab

SUMMARY:
Central serous chorioretinopathy (CSC) has been known since it was first described by Von Graefe and termed "idiopathic detachment of the macula" in 1866, is a well-characterized disorder leading to serous neurosensory elevation of the central macula. The acute form of the disease is associated with focal leakage at the level of the retinal pigment epithelium (RPE) demonstrated with fluorescein angiography (FA). The disorder is self-limited in the majority of patients, who also regain excellent vision. Occasionally, the neurosensory detachment persists and leads to pigment epithelial and photoreceptor damage with visual impairment.

The purpose of this clinical study is report the use of intravitreal bevacizumab is a new option in the treatment of the chronic or recurrent CSC.

ELIGIBILITY:
Inclusion Criteria

* Any visual acuity.
* Central serous chorioretinopathy

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2006-04 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitzy E Torres Soriano, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico